CLINICAL TRIAL: NCT03667001
Title: Comparing Analgesic Efficacy of Systemic Lidocaine Against Placebo in General Anesthesia in Bariatric Surgery: Prospective, Randomized, Double-blinded, Placebo Controlled, Mono-Center Study
Brief Title: Comparing Analgesic Efficacy of Systemic Lidocaine Against Placebo in General Anesthesia in Bariatric Surgery
Acronym: COALAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Miodrag Filipovic, Prof. Dr. med. (Other)
Responsible Party: Sponsor-Investigator, Miodrag Filipovic, Prof. Dr. med., Deputy Head of the Clinic for Anesthesiology and Intensive Care, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTU 17/026
Record Dates: First submitted 2018-08-24; First posted 2018-09-12 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Pain, Postoperative
Keywords: systemic lidocain
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: The investigators plan to evaluate the analgesic effect of systemic Lidocaine in Addition to general anesthesia during bariatric surgery.
  * Lidocaine group: perioperative application of systemic Lidocaine up to four hours from end of surgical procedures.
  * Control group: perioperative application of Placebo (NaCl 0.9%) up to four hours from end of surgical procedures.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Measures taken to minimize or avoid bias include randomization and blinding of participants after they have given their informed consent. Blinding of medical practitioner and medical personnel will be conducted by provision of equal looking and packing of IMPs, which will be fabricated individually for each patient and on request one to two days before surgery by the pharmacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine Hydrochloride (Experimental): * 1.5 mg/kg lean body mass lidocaine (lidocaine 1%) bolus I.V. as general anesthesia steady state concentration is accomplished
  * 1.5 mg/kg lean body mass/h lidocaine I.V. with beginning of surgical procedures
  * after completion of surgery: transfer to PACU, pain evaluation for 48 hours
  * duration of intervention: lidocaine infusion up to four hours from completion of surgery, or till transfer to surgical ward
  Interventions: Drug: Lidocaine Hydrochloride
- Saline Solution (Placebo Comparator): * 0.15 ml/kg lean body mass saline 0.9% bolus I.V. as general anesthesia steady state concentration is accomplished
  * 0.15 ml/kg lean body mass/h saline 0.9% I.V. with beginning of surgical procedure
  * after completion of surgery: transfer to PACU, pain evaluation for 48 hours
  * duration of intervention: saline infusion up to four hours from completion of surgery, or till transfer to surgical ward
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — The intervention to be studied will be the additional application of systemic lidocaine 1% dosed 1.5 ml/kg LBM to general anesthesia in bariatric surgery. Patients, randomly assigned to one study group, will be surveyed for 48 hours after completion of surgery, experienced pain, occurrence of PONV, time to first defecation and length of hospitalization will be monitored. Patients, medical practitioner, nurses and investigators will be blinded by utilization of equal appearance and packing of IMPs, which will be fabricated individually for each patient and on request one to two days before surgery by the pharmacy. Each patient will self-evaluate his maximal experienced pain eight-hourly during a sequence of 48 hours after completion of surgery.
  Other Names: Lidocaine Group
  Arms: Lidocaine Hydrochloride
Drug: Saline Solution — The intervention to be studied will be the additional application of NaCl 0.9% dosed 1.5 ml/kg LBM to general anesthesia in bariatric surgery as a placebo. Patients, randomly assigned to one study group, will be surveyed for 48 hours after completion of surgery, experienced pain, occurrence of PONV, time to first defecation and length of hospitalization will be monitored. Each patient will self-evaluate his maximal experienced pain eight-hourly during a sequence of 48 hours after completion of surgery.
  Other Names: Placebo Group
  Arms: Saline Solution

SUMMARY:
The investigators plan to evaluate the analgesic effect of systemic Lidocaine in addition to general anesthesia during bariatric surgery. Patients will be subdivided into a "Lidocaine group" and a "Control group".

The primary outcome will be the proportion of patients suffering from higher pain intensity within the first four hours after bariatric surgery.

Secondary outcomes include the average maximal pain intensity during first four hours and during 48 hours, total opiate consumption, occurence of postoperative nausea and vomiting, time to first defecation and total time spent in hospital.

DETAILED DESCRIPTION:
Postoperative pain is a common problem in today's surgery, although pain management techniques have improved in the last years. Systemic application of lidocaine has gained interest since several studies have shown its analgesic, anti-inflammatory and antihyperalgesic properties. In this clinical trial the analgesic effect of intravenously administrated lidocaine is compared with placebo. Despite longstanding use as an antiarrhythmic agent and its use in many clinical trial as analgesic, lidocaine is not licensed for this indication and application. Current studies, setting the focus on abdominal surgery, indicated that the systemic application of lidocaine was associated with fewer intensity of pain at rest and during mobilization and resulted in a decrease of patients'opiate consumption.

The intervention to be studied will either be the additional application of systemic lidocaine 1% to general anesthesia in bariatric surgery or the application of placebo. Patients, randomly assigned to one study group, will be surveyed for 48 hours after completion of surgery, experienced pain, occurrence of PONV, time to first defecation and length of hospitalization will be monitored. The population to be studied will include 140 patients listed for bariatric surgery at the Kantonsspital St. Gallen. Patients, medical practitioner, nurses and investigators will be blinded. Each patient will self-evaluate his maximal experienced pain eight-hourly during a sequence of 48 hours after completion of surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic bariatric surgery
* ASA classification I - III
* age 18 - 80
* given informed consent

Exclusion Criteria:

* no written consent
* allergy to the investigational product
* cardiac arrhythmia (pacemaker)
* liver dysfunction (Child-Pugh classification A, B or C)
* pregnancy
* central nervous disease
* chronic pain and pre-existing opiate prescription
* expected non-compliance
* drug/alcohol abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative VAS/NRS Score | 0 - 4 hours after surgery
  Any development of VAS/NRS score > 3 (Visual Analog Scale/Numeric Rating Scale ranging from minimum 0 to maximum 10 points, with 0 points as "no pain" to 10 points as "severe pain") , in hourly measurements within the first four hours after completion of bariatric surgery to evaluate the pain experienced by patients after the surgical intervention

SECONDARY OUTCOMES:
Average experienced maximal pain during the first four hours and 48 hours after Surgery | 0 - 48 hours after surgery
  Average experienced maximal pain during the first four hours and 48 hours (in hourly measurements on post anesthesia care unit (PACU) and in eight-hourly measurements on surgical ward) is assessed by VAS/NRS score (Visual Analog Scale/Numeric Rating Scale ranging from minimum 0 to maximum 10 points, with 0 points as "no pain" to 10 points as "severe pain").
Occurence of Postoperative Nausea and Vomiting after Surgery | 0 - 48 hours after surgery
  Any event of postoperative nausea and vomiting (PONV) (subdivided by event of no nausea (PONV = 0), event of nausea without vomiting (PONV = 1) and event of nausea with vomiting (PONV = 2)) during first 48 hours after completion of surgery
Time to first Defecation | 0 - 48 hours after surgery
  Time to first defecation (quantified in hours)
Duration of Hospitalization | 0 - 48 hours after surgery
  Duration of hospitalization (quantified in days)
Total Amount of Opiate Consumption | 0 - 48 hours after surgery
  The total amount of opiates (given during surgery and on PACU and administrated by nurse controlled analgesia on surgical ward)

CONTACTS AND LOCATIONS:
Overall Officials: Miodrag Filipovic, Prof.Dr.med., Principal Investigator — Deputy Head of the Clinic for Anesthesiology & Intensive Care
Locations (1):
- Cantonal Hospital of St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Background] McCarthy GC, Megalla SA, Habib AS. Impact of intravenous lidocaine infusion on postoperative analgesia and recovery from surgery: a systematic review of randomized controlled trials. Drugs. 2010 Jun 18;70(9):1149-63. doi: 10.2165/10898560-000000000-00000. PMID 20518581
- [Background] Vigneault L, Turgeon AF, Cote D, Lauzier F, Zarychanski R, Moore L, McIntyre LA, Nicole PC, Fergusson DA. Perioperative intravenous lidocaine infusion for postoperative pain control: a meta-analysis of randomized controlled trials. Can J Anaesth. 2011 Jan;58(1):22-37. doi: 10.1007/s12630-010-9407-0. PMID 21061107
- [Background] Cui W, Li Y, Li S, Wang R, Li J. Systemic administration of lidocaine reduces morphine requirements and postoperative pain of patients undergoing thoracic surgery after propofol-remifentanil-based anaesthesia. Eur J Anaesthesiol. 2010 Jan;27(1):41-6. doi: 10.1097/EJA.0b013e32832d5426. PMID 19478674
- [Background] Herroeder S, Pecher S, Schonherr ME, Kaulitz G, Hahnenkamp K, Friess H, Bottiger BW, Bauer H, Dijkgraaf MG, Durieux ME, Hollmann MW. Systemic lidocaine shortens length of hospital stay after colorectal surgery: a double-blinded, randomized, placebo-controlled trial. Ann Surg. 2007 Aug;246(2):192-200. doi: 10.1097/SLA.0b013e31805dac11. PMID 17667496
- [Background] Groudine SB, Fisher HA, Kaufman RP Jr, Patel MK, Wilkins LJ, Mehta SA, Lumb PD. Intravenous lidocaine speeds the return of bowel function, decreases postoperative pain, and shortens hospital stay in patients undergoing radical retropubic prostatectomy. Anesth Analg. 1998 Feb;86(2):235-9. doi: 10.1097/00000539-199802000-00003. PMID 9459225
- [Background] Weibel S, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, Eberhart LH, Poepping DM, Afshari A, Kranke P. Efficacy and safety of intravenous lidocaine for postoperative analgesia and recovery after surgery: a systematic review with trial sequential analysis. Br J Anaesth. 2016 Jun;116(6):770-83. doi: 10.1093/bja/aew101. PMID 27199310
- [Background] De Oliveira GS Jr, Duncan K, Fitzgerald P, Nader A, Gould RW, McCarthy RJ. Systemic lidocaine to improve quality of recovery after laparoscopic bariatric surgery: a randomized double-blinded placebo-controlled trial. Obes Surg. 2014 Feb;24(2):212-8. doi: 10.1007/s11695-013-1077-x. PMID 24036842
- [Background] Janmahasatian S, Duffull SB, Ash S, Ward LC, Byrne NM, Green B. Quantification of lean bodyweight. Clin Pharmacokinet. 2005;44(10):1051-65. doi: 10.2165/00003088-200544100-00004. PMID 16176118
- [Derived] Yurttas T, Djurdjevic M, Schnider TW, Filipovic M. Analgesic efficacy of systemic lidocaine using lean body mass based dosing regime versus placebo in bariatric surgery: a prospective, randomised, double-blind, placebo-controlled, single-centre study. Br J Anaesth. 2023 Jul;131(1):122-129. doi: 10.1016/j.bja.2023.03.027. Epub 2023 May 12. PMID 37183098

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT03667001/Prot_SAP_001.pdf